CLINICAL TRIAL: NCT00527059
Title: Renal Effects of Levosimendan in Patients Admitted With Acute Decompensated Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEV1068
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Heart Failure; Renal Insufficiency
Keywords: Cardiorenal syndrome
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome | interventions — Simendan; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients with acute heart failure
  Interventions: Drug: Levosimendan in addition to standard therapy
- 2 (Active Comparator): standard therapy for heart failure
  Interventions: Drug: spironolactone, beta-blockers,ecc

INTERVENTIONS:
Drug: Levosimendan in addition to standard therapy — intravenous infusion of levosimendan (10 minutes bolus with 6 mcg/Kg according to physician judgement, followed by 0.1 mcg/Kg/min for 24 hours) in addition to standard therapy
  Arms: 1
Drug: spironolactone, beta-blockers,ecc
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of levosimendan infusion, in addition to standard therapy,on renal function in patients with Acute Heart Failure,compared with standard therapy alone.

DETAILED DESCRIPTION:
The term "cardiorenal syndrome" has been applied to the presence or development of a renal dysfunction in HF patients and may be the major precipitant of decompensation and cause for admission in these patients. The renal hypoperfusion that occurs with cardiac injury can lead to sodium and water retention and activation of the renin-angiotensin-aldosterone system and neurohormonal pathways with resultant deleterious effects on the myocardium. A vicious cycle may then ensue and be associated with increased cardiovascular complications. In this regard, renal dysfunction is of a functional nature and thus means to intervene with this vicious cycle need to be sought.

Several studies already demonstrated the deleterious effects of renal dysfunction on prognosis in patients with HF due to chronic left ventricular dysfunction.

Levosimendan increases myocardial contractility without significant changes in the intracellular calcium ion and cyclic adenosine monophosphate concentrations and does not enhance myocardial oxygen demand. By its action on the potassium channels this drug also dilates the coronary and peripheral arteries and exerts an anti-ischemic,anti-stunning effect. To date, the effects of levosimendan on renal function in patients with worsening chronic HF, remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* an ejection fraction (EF) 40% by transthoracic echocardiogram,
* a baseline pulmonary capillary wedge pressure (PCWP) 20 mm Hg
* a MDRD (Modification of Diet Renal Disease) score > 30 and < 60
* and a standard therapy for HF that should include angiotensin converting enzyme inhibitors, angiotensin receptor blockers, aldosterone blocking agents (spironolactone) and beta-blockers, unless contraindicated

Exclusion Criteria:

* patients receiving other oral or i.v. inotropes,
* oral or i.v. diuretics
* or receiving nitroglycerine or nitroprusside,
* patients with systolic blood pressure <110 mmHg,
* mechanical ventilation,
* anticipated survival <30 days,
* absence of thoracic windows for echocardiography,
* acute coronary syndromes,
* sustained ventricular tachycardia or ventricular fibrillation,
* documented renal artery stenosis, requiring dialysis,
* requiring admission primarily for concurrent morbidity,
* severe aortic or mitral regurgitation,
* left ventricular failure primarily from uncorrected obstructive valvular disease, hypertrophic obstructive cardiomyopathy, restrictive/obstructive cardiomyopathy,
* uncorrected thyroid disease,
* known amyloid cardiomyopathy
* or known malfunctioning artificial heart valve.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-10; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: GFR measured by inulin Clearance. | 0, 24. 48 and 72 hours after Levosimendan infusion starting

SECONDARY OUTCOMES:
Secondary endpoints: •Other renal function measures: BUN, albumin, urine volume, sodium excretion and plasma sodium, and cystatin. •Hemodynamic parameters: PCWP, PAP, cardiac output, HR, BP, renal blood flow. | 0,1,24,48 and 72 hours after Levosimendan infusion started

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fedele, professor, Principal Investigator — Department of Cardiovascular, Respiratory and Morphological Sciences, University of Rome La Sapienza
Locations (1):
- Department of Cardiovascular, Respiratory and Morphological Sciences, University of Rome La Sapienza, Rome, Viale Del Policlinico 155, Italy

REFERENCES:
- [Derived] Fedele F, Bruno N, Brasolin B, Caira C, D'Ambrosi A, Mancone M. Levosimendan improves renal function in acute decompensated heart failure: possible underlying mechanisms. Eur J Heart Fail. 2014 Mar;16(3):281-8. doi: 10.1002/ejhf.9. Epub 2013 Dec 11. PMID 24464960